CLINICAL TRIAL: NCT03575715
Title: Endobronchial Ultrasound Image Features in the Diagnosis of Peripheral Pulmonary Lesions
Brief Title: EBUS Image Features in the Diagnosis of PPLs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Xu Lei, Chief Physician, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Chest007
Record Dates: First submitted 2018-06-21; First posted 2018-07-02 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Endobronchial Ultrasound
Keywords: endobronchial ultrasound; peripheral pulmonary lesions; image features

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EBUS group (Experimental): EBUS and guide sheath (GS) are inserted into bronchi in the assistance of navigation bronchoscopy. The EBUS probe and GS are confirmed to reach the lesion by EBUS images, cytologic and pathologic specimens are obtained with or without fluoroscopic guidance.
  Interventions: Device: EBUS

INTERVENTIONS:
Device: EBUS — EBUS is performed using an endoscope ultrasound system , which is equipped with a 20-MHz mechanical radial-type probe (UM-S20-17S;Olympus) with an external diameter of 1.4 mm and a GS (K-201; Olympus).

SUMMARY:
The study is aimed to evaluate the sensitivity, specificity, positive predictive value, negative predictive value and accuracy rate of endobronchial ultrasound (EBUS) image features in diagnosing peripheral pulmonary lesions (PPLs).

DETAILED DESCRIPTION:
The study is designed as a single center prospective trial. The participating center is Department of Ultrasound, Shanghai chest Hospital, Shanghai Jiao Tong University, China. The study is expected to enroll 200 patients. The investigator evaluates the sensitivity, specificity, positive predictive value, negative predictive value and accuracy rate of EBUS image features in diagnosing PPLs. EBUS is performed using an endoscope ultrasound system, which is equipped with a 20-MHz mechanical radial-type probe (UM-S20-17S;Olympus) with an external diameter of 1.4 mm.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are older than 18 year-old.
2. Chest CT shows PPLs suspected to be malignant that need to be confirmed by pathology. The lesion is surrounded by lung parenchyma and invisible in standard bronchoscopy.
3. Patients who agree to undergo bronchoscopy without any contraindications.
4. Patients who have good compliance and sign informed consent.

Exclusion Criteria:

1. Absence of bronchus leading to or adjacent to the lesion from CT scan.
2. Refusal of participation.
3. Severe cardiopulmonary dysfunction and other indications that can't receive bronchoscopy.
4. Presence of concomitant endobronchial lesion during the bronchoscopy procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The diagnostic value of EBUS image features | one year
  The diagnostic value includes sensitivity, specificity, positive predictive value, negative predictive value and accuracy rate.

SECONDARY OUTCOMES:
EBUS image features of adenocarcinoma | one year
  Making invasive EBUS image features of adenocarcinoma and non-invasive adenocarcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Lei Wang, MD, Principal Investigator — Shanghai Chest Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chao TY, Lie CH, Chung YH, Wang JL, Wang YH, Lin MC. Differentiating peripheral pulmonary lesions based on images of endobronchial ultrasonography. Chest. 2006 Oct;130(4):1191-7. doi: 10.1378/chest.130.4.1191. PMID 17035455
- [Background] Izumo T, Sasada S, Chavez C, Matsumoto Y, Tsuchida T. Radial endobronchial ultrasound images for ground-glass opacity pulmonary lesions. Eur Respir J. 2015 Jun;45(6):1661-8. doi: 10.1183/09031936.00167914. Epub 2015 Jan 8. PMID 25573408
- [Background] Kurimoto N, Murayama M, Yoshioka S, Nishisaka T. Analysis of the internal structure of peripheral pulmonary lesions using endobronchial ultrasonography. Chest. 2002 Dec;122(6):1887-94. doi: 10.1378/chest.122.6.1887. PMID 12475821
- [Background] Yasufuku K. Current clinical applications of endobronchial ultrasound. Expert Rev Respir Med. 2010 Aug;4(4):491-8. doi: 10.1586/ers.10.39. PMID 20658910
- [Background] Travis WD, Rekhtman N, Riley GJ, Geisinger KR, Asamura H, Brambilla E, Garg K, Hirsch FR, Noguchi M, Powell CA, Rusch VW, Scagliotti G, Yatabe Y. Pathologic diagnosis of advanced lung cancer based on small biopsies and cytology: a paradigm shift. J Thorac Oncol. 2010 Apr;5(4):411-4. doi: 10.1097/JTO.0b013e3181d57f6e. No abstract available. PMID 20357614